CLINICAL TRIAL: NCT03409016
Title: Identifying Biomarkers of Immune-Related Toxicity in Cancer Patients Treated With Immune Checkpoint Inhibitors; A Pilot Project
Brief Title: Biomarkers of Immune-Related Toxicity
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1940.cc
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Metastatic Cancer
Keywords: Immune Checkpoint Inhibitors; Biomarkers; Immune Related Adverse Event
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immune Checkpoint Inhibitor Therapy: Patients starting treatment with ipilimumab, nivolumab, pembrolizumab, or atezolizumab, alone or in combination, for treatment of a metastatic solid tumor cancer will be enrolled. Patients will receive checkpoint inhibitor therapy per standard protocol. There are no study-related medications or interventions beyond blood testing.
  Interventions: Other: Blood Testing
- Control: An additional 18 patients starting standard chemotherapy will be enrolled as a control population. Patients will receive chemotherapy per standard protocol
  Interventions: Other: Blood Testing

INTERVENTIONS:
Other: Blood Testing — Patients will undergo therapy per standard protocol. There are no study-related medications or interventions beyond blood testing.

SUMMARY:
This is a single-center, correlative pilot study evaluating potential biomarkers predictive of immune-related adverse events associated with immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
This is a single-center, correlative pilot study evaluating potential biomarkers predictive of immune-related adverse events associated with immune checkpoint inhibitor therapy. The study includes a control population of patients receiving standard chemotherapy as a comparator. Patients will undergo blood draws at 4 time-points while on standard of care treatment. There are no study-related medications or interventions beyond blood sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic solid tumor cancer of any primary site, with the exception of lymphoma
2. ≥18 years of age
3. Life expectancy >6 months
4. Starting new regimen of ipilimumab, nivolumab, pembrolizumab or atezolizumab as a single agent or in combination according to standard of care or through compassionate use granted by the pharmaceutical company (immune checkpoint inhibitor arm only) OR Starting new regimen of standard cytotoxic chemotherapy (control arm only)
5. Provision to sign and date the consent form
6. Stated willingness to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

1. Prior immune checkpoint inhibitor therapy with anti-CTLA4, anti-PD1 or anti-PD-L1 targeting agent
2. Known autoimmune disease
3. Known acute or chronic infection, including viral infections such as Hepatitis B, C, and HIV
4. Chronic treatment with immune suppressive medications, including steroids, at the time of study enrollment
5. Concomitant treatment with a monoclonal antibody in addition to cytotoxic chemotherapy (i.e. bevacizumab, cetuximab, trastuzumab) (control arm only)
6. Known pregnancy or lactation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients will be enrolled only at the University of Colorado Cancer Center in the outpatient clinic setting.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Identifying biomarkers predictive of immune-related toxicity associated with immune checkpoint inhibitor therapy. | 30 Months
  Difference in baseline inflammatory/autoimmune marker(s) in patients developing immune-related adverse events on immune checkpoint inhibitor therapy according to CTCAE v 4.0 versus those who do not

SECONDARY OUTCOMES:
Change in inflammatory/autoimmune markers. | 6 Months
  To evaluate the change in inflammatory/autoimmune markers prior to and at 3 time points on immune checkpoint inhibitor therapy, with comparison to patients treated with standard chemotherapy
Change in inflammatory/autoimmune markers | 6 months
  To evaluate the impact of change in these markers on patient reported adverse events using the PRO-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Davis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No